CLINICAL TRIAL: NCT05989763
Title: Interrogating the Pathophysiological Mechanisms of Constipation in Patients With Systemic Sclerosis
Acronym: TEA in SSc
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Principal Investigator, Zsuzsanna Hortobagyi Mcmahan, Associate Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HSC-MS-23-0531; 1R01AR081382-01A1 (NIH)
Record Dates: First submitted 2023-08-04; First posted 2023-08-14 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Systemic Sclerosis; Constipation; Gastrointestinal Motility Disorder; Autonomic Dysfunction
MeSH Terms: conditions — Scleroderma, Systemic; Constipation; Primary Dysautonomias

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Transcutaneous Electrical Acustimulation (TEA) (Experimental)
  Interventions: Device: Transcutaneous Electrical Acustimulation (TEA)
- Sham-TEA (Sham Comparator)
  Interventions: Device: Sham-TEA

INTERVENTIONS:
Device: Transcutaneous Electrical Acustimulation (TEA) — TEA will then be administrated for 1 hour twice daily for a period of 4 weeks
  Arms: Transcutaneous Electrical Acustimulation (TEA)
Device: Sham-TEA — Sham TEA will then be administrated for 1 hour twice daily for a period of 4 weeks
  Arms: Sham-TEA

SUMMARY:
The purpose of this study is to determine whether transcutaneous electrical acustimulation (TEA) alters systemic sclerosis (SSc)-related colonic and anorectal physiology by enhancing autonomic nervous system (ANS) function. The study will examine the effects of TEA on slow colonic transit (SCT) and rectal hyposensitivity (RH), to examine whether TEA improves autonomic dysfunction and modulates inflammatory pathways.

ELIGIBILITY:
Inclusion Criteria

* Patients with SSc-constipation from Aim 1 of the study
* Patients with SCT (>20% radiopaque marks left in the colon 5 days (120 hours) after swallowing the Sitzmark capsule or patients with RH (defined in Aim 1)
* Patients not yet on therapy for constipation or patients who continue to experience constipation while on stable therapy for one month prior to TEA.

Exclusion Criteria

-Patients with symptoms of both diarrhea and constipation but not predominantly symptoms of constipation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-02-17 (Actual); Primary Completion 2028-08-14 (Estimated); Study Completion 2029-09-01 (Estimated)

PRIMARY OUTCOMES:
Change in slow colonic transit (SCT) | baseline, week 4 (visit 2)
  slow colonic transit (SCT) is defined by more than 5 (20%) of Sitz markers retained 5 days after ingestion

SECONDARY OUTCOMES:
Change in rectal hyposensitivity as assessed by the anorectal manometry | baseline, week 4 (visit 2)
Change in autonomic dysfunction as assessed by the Heart rate variability (HRV) measures | baseline, week 4 (visit 2)
Change in autonomic dysfunction as assessed by the COMPASS-31 measures | baseline, week 4 (visit 2)
  This is a 31 item questionnaire and scores range from 0-100 a higher score indicating more severe autonomic dysfunction
Change in inflammatory cytokines (IL-6, Tumour Necrosis Factor alpha (TNF-alpha) ), | baseline, week 4 (visit 2)

CONTACTS AND LOCATIONS:
Overall Officials: Zsuzsanna H McMahan, MD, MHS (M-PI), Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No